CLINICAL TRIAL: NCT00813085
Title: A Randomized Trial of Electronic Integration of Care for Better Diabetes Outcomes; The COMPETE II Study
Acronym: COMPETEII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Health Canada (Other Government)
Responsible Party: Anne M Holbrook, PharmD, MD, MSc, St Joseph's Healthcare
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 02-2068
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2008-12-22 (Estimated); Status verified 2008-12

CONDITIONS: Diabetes
Keywords: Diabetes; Computerized clinical decision support; shared care; patient self-monitoring; quality of care; complex interventions; composite outcomes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic disease management decision support (Other): An electronic Diabetes Tracker embedded in a Core Data Set (DT/CDS) supported by an automated telephone reminder system (ATRS).
  Interventions: Other: Electronic disease management decision support
- 2 (No Intervention): Usual care by Family Physician

INTERVENTIONS:
Other: Electronic disease management decision support — A Diabetes Tracker embedded in a Core Data Set (DT/CDS) supported by an automated telephone reminder system (ATRS)
  Other Names: Intervention
  Arms: Electronic disease management decision support

SUMMARY:
This study will evaluate whether the use of an electronic diabetes tracker by both patients and family physicians in Ontario improves diabetes outcomes, satisfaction with care and with technology and health data privacy issues. As part of the study, the investigators will be able to test whether practices that use computers perform any better than practices using paper. The investigators also will be developing the first Canadian computerized chart summary for each patient that can be communicated securely in emergencies (the Emergency Health Record) and read by all current electronic systems.

ELIGIBILITY:
Inclusion Criteria:

* Adult, cognitively intact, consenting people with diabetes within enrolled practices

Exclusion Criteria:

* Non-english speaking
* Cognitively impaired

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2002-04; Primary Completion 2003-09 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Comparison of change in diabetes quality of care between intervention and usual care group. | 6 months follow-up

SECONDARY OUTCOMES:
Change in diabetes risk factor variables, satisfaction with care and technology, quality of life and health care utilization, health data privacy issues. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Holbrook, MD,PharmD,MSc, Principal Investigator — McMaster University
Locations (1):
- St Joseph's Healthcare & Mcmaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Holbrook A, Thabane L, Keshavjee K, Dolovich L, Bernstein B, Chan D, Troyan S, Foster G, Gerstein H; COMPETE II Investigators. Individualized electronic decision support and reminders to improve diabetes care in the community: COMPETE II randomized trial. CMAJ. 2009 Jul 7;181(1-2):37-44. doi: 10.1503/cmaj.081272. PMID 19581618
- See also: COMPETE group website for all series of Compete trials and work — http://www.compete-study.com